CLINICAL TRIAL: NCT03886038
Title: The Immunogenicity and Efficacy of Subunit Vaccine Against Herpes Zoster in RA Treated With JAK-inhibitors (VACCIMIL-ZOSTER)
Brief Title: Subunit Vaccine Against Herpes Zoster in RA Patients Treated With JAK-inhibitors (VACCIMIL-ZOSTER)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VACCIMIL-ZOSTER
Record Dates: First submitted 2019-01-02; First posted 2019-03-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Arthritis; Healthy Controls
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RA patients on JAK inhibitors (Active Comparator): RA patients treated with JAK inhibitors as a monotherapy or in combination with methotrexate/other DMARDs/prednisone for at least 3 months will receive two doses of Shingrix vaccine administrated with at least 2 months apart
  Interventions: Biological: Shingrix
- healthy controls (Active Comparator): healthy individuals without any rheumatic disease or not treated with any immunosupressive drug for any other condition will receive two doses of Shingrix vaccine administrated with at least 2 months apart
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: Shingrix — immunization with 2 doses of a subunit vaccine against herpes-zoster (Shingrix) administrated with at least 2 months apart

SUMMARY:
Background. A new subunit vaccine against herpes zoster (HZ) has recently been approved for vaccination of adults i in Sweden. This vaccine (Shingrix) elicits a strong cellular and humoral immune response in healthy adults regardless of age. Studies on the immunogenicity and efficacy of this vaccine in immunosuppressed patients, such as patients with rheumatoid arthritis (RA), are scarce.

Objectives. To investigate: 1) the immunogenicity of subunit vaccine against HZ in patients with RA treated with janus kinase (JAK)-inhibitors compared to healthy controls; 2) the tolerability of subunit vaccine against HZ 3) long-term immunogenicity of two doses of subunit HZ vaccine 4) the impact of smoking habits and alcohol consumption on the immunogenicity of vaccine and protection against HZ 5) the efficacy of this vaccine.

Methodology. Patients with RA, regularly followed at the Skåne University Hospital, section for rheumatology in southern Sweden are eligible for the study and will be offered vaccination. Blood samples will be collected immediately before the first vaccine dose and 4-6 weeks after the second dose and thereafter 3 and 5 years after the second vaccination. The levels of antibodies to glycoprotein E (gE) will be measured with standard ELISA on the blood samples collected at vaccination, 4-6 weeks following the second vaccination and after 3 and 5 years. A flow-cytometric assay will be used for the detection of the cell-mediated immunity (number of antigen specific CD4+ T-cells) against the varicella-zoster virus. The prevalence of HZ among patients participating in the study will be compared to in-patient and out-patient registry data on the corresponding infections among age- and sex- matched non-vaccinated controls using data from the regional health and care registry in southern Sweden.

DETAILED DESCRIPTION:
Background. Treatment with JAK-inhibitors has been shown to improve the signs and symptoms of rheumatoid arthritis (RA) and delay the development of radiographic damage. However, these remedies have been shown to increase risk of herpes zoster (HZ) infections in RA. Currently available live attenuated vaccine against HZ is contraindicated in patients receiving immunosuppressive treatments. A new subunit vaccine against HZ has recently been approved for vaccination of adults in Sweden. This vaccine (Shingrix) has been shown to elicit a strong cellular and humoral immune response in healthy adults regardless of age. Studies on the immunogenicity and efficacy of this vaccine in immunosuppressed patients, such as patients with RA, are scarce.

Objectives. To investigate: 1) the immunogenicity of 2 doses of HZ vaccine (Shingrix) administrated at least 2 months apart in patients with RA treated with JAK-inhibitors for at least 3 months compared to immunogenicity of the vaccine given to healthy controls; 2) the tolerability of subunit vaccine against HZ i.e. whether vaccination is associated with increased disease activity, flare of RA or the onset of other autoimmune disease 3) long-term immunogenicity of two doses of the subunit vaccine against HZ; 4) the impact of smoking habits and alcohol consumption on the immunogenicity of vaccine and protection against HZ infection 5) the efficacy of the vaccine in preventing HZ.

Methodology. Patients with RA, regularly followed at the Skåne University Hospital, section for rheumatology already treated with JAK inhibitors for at least 3 months are eligible for the study and will be offered to participate in the study. At vaccination, the clinical examination is performed, and data on disease and treatment characteristics, co-morbidity, smoking and alcohol habits are collected. All participants are encouraged to take the notice of changes in the existing RA or other unexpected side effects following vaccinations. Blood samples will be collected immediately before the first vaccination and 4-6 weeks after the second dose of the vaccine and thereafter 3 and 5 years after vaccination. The levels of antibodies to glycoprotein E (gE) using standard ELISA will be performed on the blood samples collected at vaccination, 4-6 weeks following the second dose of the vaccine and after 3 and 5 years. A flow-cytometric assay will be used for the detection of the cell-mediated immunity (number of antigen specific CD4+ T-cells) against the varicella-zoster virus. The prevalence of HZ among patients participating in the study will be compared to in-patient and out-patient register data on the corresponding infections among age- and sex- matched non-vaccinated controls using data from the regional health and care registry in the Skåne region, southern Sweden.

Impact. Results from this project will provide the evidence whether 2 doses of the subunit HZ vaccine is immunogenic, safe and efficacious in patients with RA treated with JAK- inhibitors and which factors can influence the efficacy of the vaccine. These results can be used for the future recommendations on vaccination against HZ and when in relation to treatment the immunization should be performed in order to reach the best protection. In the long term this should result in decreased morbidity in HZ infections, complication of those infections and lower health-care costs.

ELIGIBILITY:
Inclusion Criteria:

age>18 years RA diagnosis RA patients treated with JAK-inhibitors as monotherapy or in combination with MTX and/or other DMARDs/prednisolone for at least 3 months (group1) regulary follow up at the rheumatology departmenet

Exclusion Criteria:

* pregnancy
* breastfeeding
* allergi against some of compnents in the vaccine
* ongoing infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
the differences in serological response between the groups | 4-6 week after two vaccine doses
  levels of antibodies to glycoprotein E (gE)
the differences in the T cells response between the groups | 4-6 week after two vaccine doses
  number of antigen specific CD4+ T-cells in blood samples collected at vaccination and after the second vaccine dose

SECONDARY OUTCOMES:
the differences in antibody levels to glycoprotein E between the groups 3 and 5 after vaccination | up to 5 years after vaccination
  levels of antibodies to glycoprotein E (gE) measured in blood samples taken 3 and 5 years after the second vaccine dose

OTHER OUTCOMES:
the number of HZ infections registerd among patricipants in the study compared to non-vaccinated controls | up to 5 years after vaccination
  the occurrence of HZ infections among patients participating in the study compared to age- and sex- matched non-vaccinated population from the same geographic area

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University hospital, Dept of rheumatology, Lund, Sweden

REFERENCES:
- [Derived] Kallmark H, Gullstrand B, Kahn F, Grenmyr E, Kahn R, Einarsson JT, Bengtsson AA, Kapetanovic MC. Impaired cellular immune responses to herpes zoster subunit vaccine in patients with rheumatoid arthritis receiving Janus kinase inhibitors. Rheumatology (Oxford). 2026 Jan 8;65(1):keaf626. doi: 10.1093/rheumatology/keaf626. PMID 41330694
- [Derived] Kallmark H, Bergstrom T, Nagel J, Gullstrand B, Einarsson JT, Bengtsson AA, Kapetanovic MC. Serologic immunogenicity and safety of herpes zoster subunit vaccine in patients with rheumatoid arthritis receiving Janus kinase inhibitors. Rheumatology (Oxford). 2024 Jul 1;63(7):2024-2033. doi: 10.1093/rheumatology/kead552. PMID 37851412